CLINICAL TRIAL: NCT06344273
Title: The Effect of Lower Extremity ROM Exercises on Hypotension, Fatigue and Hemodialysis Comfort in Individuals Receiving Hemodialysis Treatment
Brief Title: The Effect of Lower Extremity ROM Exercises on Hypotension, Fatigue, and Hemodialysis Comfort in Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Burcu01
Record Dates: First submitted 2023-07-31; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-08

CONDITIONS: Hemodialysis
Keywords: fatique; hypotansion; hemodialysis comfort

STUDY DESIGN:
Intervention Model Description: The patients will be divided into the intervention group (n=32) in which 20 minutes of ROM exercise was applied and the control group (n=32) in which routine nursing care was given. For the sample calculation of the study, G power analysis was performed, type 1 error was 0.05; type 2 error 0.20; With a power of 0.80, a minimum sample size of 64 people for the experimental and control groups. The case group will be given lower extremity ROM exercises for a total of two weeks. Each individual in the case group will have lower extremity ROM exercises, each of which will last 20 minutes, at the beginning of the session and at the beginning of the hour until the end of the session. "Piper's Fatigue Scale" and Hemodialysis Comfort Scale" in the data collection form will be applied again at the end of the 1st and 2nd weeks after the sessions have started. The vital signs of the individual will be followed and recorded at each session.
Who Masked: Participant
Masking Description: You are completely free to participate in the research or not. Not participating in this research will certainly not affect the service you receive. You have the right to withdraw from the study at any time by giving notice; you may also be excluded from the study by the investigator, if deemed necessary, provided that no harm is done to your medical condition.
  If you participate in the research, you will not be charged or paid any fees for the expenses to be made in the study. In addition, at the end of the research, your information will only serve scientific purposes without revealing your identity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Lower Extremity ROM exercise will be performed for 20 minutes each at the beginning of the hour until the end of each eye session, examination and session in the case visits. "Piper's Fatigue Scale" and Hemodialysis Comfort Scale", which are part of data collection, will be applied again at the end of the 1st and 2nd week after the sessions begin. The individual's life segments will be tracked and recorded at each session.
  Interventions: Behavioral: ROM exercises
- Control Group (No Intervention): During the implementation period of the study, routine nursing care service will be provided to the patients in the control group and no additional nursing intervention will be applied. "Piper's Fatigue Scale" and Hemodialysis Comfort Scale", which are part of data collection, will be applied again at the end of the 1st and 2nd week after the sessions begin. The individual's life segments will be tracked and recorded at each session.

INTERVENTIONS:
Behavioral: ROM exercises — Each individual in the case group will have lower extremity ROM exercises, each of which will last 20 minutes, at the beginning of the session and at the beginning of the hour until the end of the session.
  Arms: experimental group

SUMMARY:
Range of motion (ROM) is a term used to describe the amount of motion in each joint in our body. Every joint in the body has a normal range of motion. Maintaining the normal opening of the joints is achieved through movement. ROM exercises reduce contractures and are very important in terms of helping to preserve muscle movements. ROM exercises are an inexpensive method that can be applied in any environment, either as a group or individually, covering all muscle-joint groups. Individuals with disabilities can perform ROM exercises individually or receive support from healthcare professionals. It provides support to venous return by increasing muscle strength in patients who are immobilized for a long time.

Based on this information, the aim of our study is to investigate the effect of lower extremity ROM exercises during hemodialysis on hypotension, fatigue and hemodialysis comfort.

The patients will be divided into the intervention group (n=32) in which 20 minutes of ROM exercise was applied and the control group (n=32) in which routine nursing care was given. For the sample calculation of the study, G power analysis was performed, type 1 error was 0.05; type 2 error 0.20; With a power of 0.80, a minimum sample size of 64 people for the experimental and control groups. The case group will be given lower extremity ROM exercises for a total of two weeks. Each individual in the case group will have lower extremity ROM exercises, each of which will last 20 minutes, at the beginning of the session and at the beginning of the hour until the end of the session. "Piper's Fatigue Scale" and Hemodialysis Comfort Scale" in the data collection form will be applied again at the end of the 1st and 2nd weeks after the sessions have started. The vital signs of the individual will be followed and recorded at each session.

DETAILED DESCRIPTION:
Chronic kidney failure (CKD) is an important disease that disrupts the fluid and electrolyte balance of the individual, hinders the execution of the body's metabolic activities, and has an increasing prevalence in the world and in our country. Waste and toxic products that cannot be disposed of because CRF disrupts homeostasis are removed from the body by hemodialysis, which is a renal replacement therapy. During the hemodialysis treatment process, individuals may encounter many physical or psychological problems that affect their quality of life such as hypotension, pain, muscle cramps, nausea, vomiting, dry skin, itching, sleep problems, fatigue, constipation, diarrhea, emotional and sexual problems.

In hemodialysis patients, various complications occur before, during and after dialysis treatment, usually within 1-4 hours. One of the most common complications during hemodialysis (intradialytic) is hypotension. The Renal Disease Outcomes Quality Initiative (KDOQI) and European Best Practice Guidelines (EBPG) define intradialytic hypotension as the development of clinical symptoms (cramp, nausea, vomiting, dizziness, discomfort…) with a decrease in systolic blood pressure of ≥20 mmHg or a decrease in mean blood pressure of >10 mmHg, and the need for nursing interventions.

Normal responses are often impaired in hemodialysis patients due to comorbidities such as cardiac dysfunction and autonomic neuropathy. Besides cardiac factors, the vascular reaction to the decrease in blood volume may also be impaired during dialysis treatment. Decreased arteriolar contraction compromises the physiological increase in systemic vascular resistance during hypovolemia. Reduction in passive and active narrowing of venules and veins reduces the shunt of blood to the central circulation and impairs venous return.

Fatigue, defined as a subjective weakness, lack of energy, is a common symptom after hemodialysis. Psychological factors such as ultrafiltration, diffusion, osmotic imbalance, changes in blood pressure, blood membrane interactions, prolonged positioning during dialysis, higher tumor necrosis factor levels, and depression all play a role in the pathogenesis of post-dialysis fatigue.

Studies have shown that physical exercise improves the exercise-functional capacity, muscle strength and quality of life of patients receiving dialysis treatment, provides blood pressure control, reduces the risk of diabetes development and cardiovascular disease, alleviates depression and anxiety symptoms, increases survival and dialysis efficiency.

Range of motion (ROM) is a term used to describe the amount of motion in each joint in our body. Every joint in the body has a normal range of motion. Maintaining the normal opening of the joints is achieved through movement. ROM exercises reduce contractures and are very important in terms of helping to preserve muscle movements. ROM exercises are an inexpensive method that can be applied in any environment, either as a group or individually, covering all muscle-joint groups. Individuals with disabilities can perform ROM exercises individually or receive support from healthcare professionals. It provides support to venous return by increasing muscle strength in patients who are immobilized for a long time.

Based on this information, the aim of our study is to investigate the effect of lower extremity ROM exercises during hemodialysis on hypotension, fatigue and hemodialysis comfort. The research was designed as a randomized controlled experimental study. The sample of the study will be included individuals who received treatment at the Private Vital Dialysis Center between July and August 2023, agreed to participate in the study and received written permission, were older than 18 years old, were open to communication, were fully oriented, could speak and understand Turkish, received hemodialysis treatment 3 times a week for 6 months or longer, did not have fistulas, did not have any conditions such as loss of sensation in their hands and lower extremities, masses, fractures and ingrown nails. Patients who do not want to participate in the study and who want to leave the research during the research process will be excluded from the study. Confidentiality of information and the aims of the study will be explained to each participant before the study, and written and verbal consent will be obtained from individuals who agree to participate in the study. Participants will be randomly assigned to either the case group or the control group. Protocol numbers will be used to randomize participants in each group. Patients with an odd number of protocol numbers will form the experimental group, and patients with an even number of protocol numbers will form the control group. The data collection form developed by the researchers as a result of the literature review related to the research will be filled before the application. The data collection form consists of the "Patient Diagnosis Form", which includes questions about sociodemographic characteristics and the disease in the first part, and "Piper's Fatigue Scale" and Hemodialysis Comfort Scale in the second part.

The patients will be divided into the intervention group (n=32) in which 20 minutes of ROM exercise was applied and the control group (n=32) in which routine nursing care was given. For the sample calculation of the study, G power analysis was performed, type 1 error was 0.05; type 2 error 0.20; With a power of 0.80, a minimum sample size of 64 people for the experimental and control groups. The case group will be given lower extremity ROM exercises for a total of two weeks. Each individual in the case group will have lower extremity ROM exercises, each of which will last 20 minutes, at the beginning of the session and at the beginning of the hour until the end of the session. "Piper's Fatigue Scale" and Hemodialysis Comfort Scale" in the data collection form will be applied again at the end of the 1st and 2nd weeks after the sessions have started. The vital signs of the individual will be followed and recorded at each session.

ELIGIBILITY:
Inclusion Criteria:

18 years and older

* Agreeing to participate in the study and receiving written consent
* Without any cognitive, sensory and mental disorders
* Able to speak and communicate in Turkish
* Place, time and person orientation
* Those who do not have sensory and motor loss in their lower extremities (plegia, parasite, etc.)
* Individuals who do not have conditions such as mass, loss of sensation, fracture, wound, lesion in the lower extremities

Exclusion Criteria:

* Refused to participate in the study
* Patients with problems such as skin infections, thrombosis, phlebitis, fractures, circulatory disorders
* Patients who have undergone pharmacological or non-pharmacological interventions that will affect their vital signs
* Patients who want to withdraw from the research will not be included in the research process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
follow-up form | 2 weeks
  the form is based on literature and created by researcher to follow patient' blood pressure. The data will enroll manually by researher on the form.
Piper Fatigue Scale | 2 weeks
  the scale consists of a total of 22 items and evaluates the patient's subjective perception of fatigue with four subscales. These are: the behavior/severity subscale assessing the impact and severity of fatigue on daily life activities (6 items; 2-7); the affective subscale covering the emotional significance attributed to fatigue (5 items; 8-12); the sensory subscale reflecting the physical, emotional, and sensory symptoms of fatigue (5 items; 13-17); and the cognitive/mental subscale reflecting the level of impact of fatigue on cognitive functions and mental state (6 items; 18-23).
  Scoring of the Scale: Subscale scores are obtained by summing the scores of all items in that subscale and dividing by the number of items. Responses for each item are evaluated on a scale of 0-10 points. The total fatigue score is obtained by summing the scores of the 22 items and dividing by the number of items. Higher scores obtained from the scale indicate a higher perceived level of fatigue.
comfort condition | 2 weeks
  we considered patients who are in both group with Hemodialysis Comfort Scale. the questionnaire is included 9 questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No